CLINICAL TRIAL: NCT06577727
Title: A Study to Collect Data to Build Artificial Intelligence Derived Algorithms for Estimating Iron Status of Children (FERROUS 2)
Brief Title: A Study to Collect Data to Build Artificial Intelligence Derived Algorithms for Estimating Iron Status of Children
Acronym: FERROUS 2
Status: Completed | Type: Observational
Sponsor: Danone Asia Pacific Holdings Pte, Ltd. (Industry)
Collaborators: KK Women's and Children's Hospital (Other Government); Srinagarind Hospital, Khon Kaen University (Other)
Responsible Party: Sponsor
Other Study IDs: EBB19GC28473 - A
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Iron Deficiency
Keywords: Algorithm; Artificial Intelligence; Iron Deficiency; IDA; Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children aged 6-72 months of age: Approximately 250 children aged above 6 months old and below 6 years of age across potential study sites.
  Subjects will be grouped by haemoglobin (Hb) level ranging from <6 g/dL to ≥ 14.0 g/dL. There will be a minimum of 10 subjects and a maximum of 25 subjects for each group.
  Interventions: Other: Gold standard blood test; Other: Imaging and videography of anatomical sites

INTERVENTIONS:
Other: Gold standard blood test — Blood test will measure haemoglobin and other parameters
Other: Imaging and videography of anatomical sites — Images and videos of anatomical sites will be collected for AI to estimate iron status

SUMMARY:
An exploratory study to collect data to build artificial intelligence derived algorithms for estimating iron status in children

DETAILED DESCRIPTION:
This is an exploratory, observational, pilot study that aims to build and measure the accuracy of an algorithm that estimates a child's iron status using images and/or videos, against gold standard venous blood sampling. Images and/or videos will be collected by healthcare professionals, together with blood test results. This data will be used to evaluate the accuracy of the algorithm and to explore potential improvements. Data on the acceptance and experience of the using the algorithm will be collected for improvements.

ELIGIBILITY:
Inclusion Criteria:

1. Children above 6 months of age and below 6 years of age
2. Written consent from parent(s) or legally acceptable representative(s), who themselves are aged ≥ 21 years old, to consent and comply with the terms and conditions of the study
3. Parent(s) should have access to the internet and a smartphone or tablet to complete study questionnaires
4. Parent(s) should be able to comprehend the content of the study and complete the study questionnaires
5. Parents(s) must be comfortable with their child having blood draws
6. Subject has a Hb level corresponding to a Hb group with open slots for participation

Exclusion Criteria:

1. Children with any medical condition that in the opinion of the investigator would not be suitable for enrolment.
2. Children with nail bed obstructions, nail polish, nails discolouration (e.g., leukonychia, melanonychia, bruising, etc.), or scarring of the lips, pigmentations on lips for thyroid dysfunction (e.g., Puettz-jeghers syndrome).
3. Children who are unable to cooperate with study procedures.
4. Employees and/or children/family members or relatives of employees of Danone Global Research & Innovation Center or the participating sites.

Ages: 6 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children between 6 to 72 months of age
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Iron AI in a clinic setting | 1 day
  Accuracy of the Iron Ai in a clinic setting, derived from:
  1. The Iron AI prediction from images/videos collected
  2. The gold standard blood test results

SECONDARY OUTCOMES:
Parental acceptability of the Iron AI | 1 day
  Parental acceptability of the Iron AI assessed via the study questionnaire [Accuracy, Usefulness, Frequency of usage, Data sharing]
Investigator's (or delegates) acceptability of Iron AI | 1 day
  Investigators (or delegates) likelihood of using the Iron AI assessed via the study questionnaire [Ease of taking images/videos, accuracy, frequency of use, recommendation to parents]

OTHER OUTCOMES:
Correlation of proposed scoring system for iron status assessment questionnaire against the gold standard blood test result | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Poh Choo Dr Khoo, Principal Investigator — KK Women's and Children's Hospital; Assoc.Prof. Suchaorn Saengnipanthkul, Principal Investigator — Srinagarind Hospital, Khon Kaen University, Khon Kaen
Locations (2):
- KK Women's and Children's Hopsital, Singapore, Singapore
- Srinagarind Hospital, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baker RD, Greer FR; Committee on Nutrition American Academy of Pediatrics. Diagnosis and prevention of iron deficiency and iron-deficiency anemia in infants and young children (0-3 years of age). Pediatrics. 2010 Nov;126(5):1040-50. doi: 10.1542/peds.2010-2576. Epub 2010 Oct 5. PMID 20923825
- [Background] Lopez A, Cacoub P, Macdougall IC, Peyrin-Biroulet L. Iron deficiency anaemia. Lancet. 2016 Feb 27;387(10021):907-16. doi: 10.1016/S0140-6736(15)60865-0. Epub 2015 Aug 24. PMID 26314490
- [Background] Khedr E, Hamed SA, Elbeih E, El-Shereef H, Ahmad Y, Ahmed S. Iron states and cognitive abilities in young adults: neuropsychological and neurophysiological assessment. Eur Arch Psychiatry Clin Neurosci. 2008 Dec;258(8):489-96. doi: 10.1007/s00406-008-0822-y. Epub 2008 Jun 20. PMID 18574611
- [Background] WHO (2008) Worldwide prevalence of anaemia 1993-2005. In: de Benoist B, McLean E, Egli I, Cogswell M, editors. WHO global database on anaemia. Geneva: World Health Organization.
- [Background] WHO (2001) Iron deficiency anaemia. Assessment, prevention, and control. A guide for programme managers. Geneva: World Health Organization.
- [Background] Anaemia in women and children (2021). World Health Organization. https://www.who.int/data/gho/data/themes/topics/anaemia_in_women_and_children?utm_content=buffer85683&utm
- [Background] Saarinen UM, Siimes MA, Dallman PR. Iron absorption in infants: high bioavailability of breast milk iron as indicated by the extrinsic tag method of iron absorption and by the concentration of serum ferritin. J Pediatr. 1977 Jul;91(1):36-9. doi: 10.1016/s0022-3476(77)80439-3. PMID 577504
- [Background] da Silva Lopes K, Yamaji N, Rahman MO, Suto M, Takemoto Y, Garcia-Casal MN, Ota E. Nutrition-specific interventions for preventing and controlling anaemia throughout the life cycle: an overview of systematic reviews. Cochrane Database Syst Rev. 2021 Sep 26;9(9):CD013092. doi: 10.1002/14651858.CD013092.pub2. PMID 34564844
- [Background] Tounian P, Chouraqui JP. [Iron in nutrition]. Arch Pediatr. 2017 May;24(5S):5S23-5S31. doi: 10.1016/S0929-693X(17)24006-8. French. PMID 28622779
- [Background] Vitamin and mineral requirements in human nutrition, Second edition, World Health Organization and Food and Agriculture Organization of the United Nations, 2004.
- [Background] Camaschella C. Iron-deficiency anemia. N Engl J Med. 2015 May 7;372(19):1832-43. doi: 10.1056/NEJMra1401038. No abstract available. PMID 25946282
- [Background] Kohli-Kumar M. Screening for anemia in children: AAP recommendations--a critique. Pediatrics. 2001 Sep;108(3):E56. doi: 10.1542/peds.108.3.e56. PMID 11533374